CLINICAL TRIAL: NCT05355857
Title: Creation of a Probabilistic Atlas of Normal Cerebral Uptake of 18F-FDG in PET/MRI.
Acronym: ATLATEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: ICube Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-008
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Brain Diseases
Keywords: FDG PET; PET-MRI; atlas; brain
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FDG injection (Other): Health volunteers with 18-F-FDG injection
  Interventions: Diagnostic Test: brain PET-MRI with 18F-FDG

INTERVENTIONS:
Diagnostic Test: brain PET-MRI with 18F-FDG — Realisation of a brain PET-MRI with 18F-FDG in 39 healthy volunteers

SUMMARY:
With 18F-FDG PET, we have few atlases of normality allowing the realization of objective quantitative analyses. An atlas of normality is a probabilistic atlas of normal FDG uptake from a representative set of brain PET images of healthy subjects. This type of atlas is essential for intra- and inter-individual comparisons.

Accurate quantitative analysis of brain 18F-FDG PET images acquired on a hybrid PET system has been shown to require an institutional normal database for statistical analyzes (Akdemir et al., JNM 2017 and Della Rosa et al Neuroinformatics, 2014).

DETAILED DESCRIPTION:
This is a prospective, monocentric, non-randomized study, with no direct individual benefit since it involved healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 20 to 50
* Absence of any history or cardiovascular, neurological or psychiatric deficit
* Signed the informed consent

Exclusion Criteria:

* Contraindication to the realization of an MRI or PET and to the injection of 18F-FDG
* People using a pacemaker or insulin pump
* People wearing a metal prosthesis or an intracerebral clip
* People with intraocular metal splinters
* People with a pathology considered incompatible for the production of the atlas according to the investigator
* Pregnant women and breastfeeding women
* Subject in period of exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Creation, from a representative set of brain PET-MRI images of healthy subjects, of a probabilistic atlas of normal FDG uptake in healthy volunteers | 30 minutes after 18F-FDG injection
  Evaluation of tracer activity at the cerebral level on the acquisition images

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided